CLINICAL TRIAL: NCT02493764
Title: A Phase III, Randomized, Double-Blind, Active Comparator-Controlled Clinical Trial to Study the Safety, Tolerability, and Efficacy of Imipenem/Cilastatin/Relebactam (MK-7655A) Versus Piperacillin/Tazobactam in Subjects With Hospital-Acquired Bacterial Pneumonia or Ventilator-Associated Bacterial Pneumonia
Brief Title: Imipenem/Relebactam/Cilastatin Versus Piperacillin/Tazobactam for Treatment of Participants With Bacterial Pneumonia (MK-7655A-014)
Acronym: RESTORE-IMI 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7655A-014; 2015-000246-34 (EudraCT Number); 163240 (Registry Identifier: JAPIC-CTI); MK-7655A-014 (Other: Merck Protocol Number)
Record Dates: First submitted 2015-07-07; First posted 2015-07-09 (Estimated); Results first posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-03

CONDITIONS: Bacterial Pneumonia
MeSH Terms: conditions — Pneumonia, Bacterial | interventions — Imipenem; relebactam; Cilastatin; Piperacillin; Tazobactam; Linezolid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMI/REL (Experimental): Imipenem 500 mg + relebactam 250 mg + cilastatin 500 mg as a FDC administered intravenously (IV) every 6 hours for a minimum of 7 days, up to 14 days. At study entry open label linezolid 600 mg will also be administered by IV every 12 hours for up to 14 days.
  Interventions: Drug: Imipenem; Drug: Relebactam; Drug: Cilastatin; Drug: Linezolid
- PIP/TAZ (Active Comparator): Piperacillin 4000 mg + tazobactam 500 mg as a FDC administered IV every 6 hours for a minimum of 7 days, up to 14 days. At study entry open label linezolid 600 mg will also be administered by IV every 12 hours for up to 14 days.
  Interventions: Drug: Piperacillin; Drug: Tazobactam; Drug: Linezolid

INTERVENTIONS:
Drug: Imipenem — Imipenem 500 mg as part of a FDC administered by IV every 6 hours for a minimum of 7 days, up to 14 days
  Arms: IMI/REL
Drug: Relebactam — Relebactam 250 mg as part of a FDC administered by IV every 6 hours for a minimum of 7 days, up to 14 days
  Arms: IMI/REL
Drug: Cilastatin — Cilastatin 500 mg as part of a FDC administered by IV every 6 hours for a minimum of 7 days, up to 14 days
  Arms: IMI/REL
Drug: Piperacillin — Piperacillin 4000 mg as part of a FDC administered by IV every 6 hours for a minimum of 7 days, up to 14 days
  Arms: PIP/TAZ
Drug: Tazobactam — Tazobactam 500 mg as part of a FDC administered by IV every 6 hours for a minimum of 7 days, up to 14 days
  Arms: PIP/TAZ
Drug: Linezolid — Linezolid 600 mg administered open-label by IV every 12 hours for up to 14 days

SUMMARY:
This study aims to compare treatment with a fixed-dose combination (FDC) of imipenem/relebactam/cilastatin (IMI/REL) with a FDC of piperacillin/tazobactam (PIP/TAZ) in participants with hospital-acquired or ventilator-associated bacterial pneumonia (HABP or VAPB, respectively). The primary hypothesis is that IMI/REL is non-inferior to PIP/TAZ in the incidence rate of all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* Requires treatment with IV antibiotic therapy for hospital-acquired bacterial pneumonia (HABP) or ventilator-associated bacterial pneumonia (VABP)
* Fulfills clinical and radiographic criteria, with onset of criteria occurring after more than 48 hours of hospitalization or within 7 days after discharge from a hospital (for HABP); or at least 48 hours after mechanical ventilation (for VABP)
* Has an adequate baseline lower respiratory tract specimen obtained for Gram stain and culture
* Has an infection known or thought to be caused by microorganisms susceptible to the IV study therapy
* Agrees to allow any bacterial isolates obtained from protocol-required specimens related to the current infection to be provided to the Central Microbiology Reference Laboratory for study-related microbiological testing, long term storage, and other future testing
* Is not of reproductive potential; or if of reproductive potential agrees to avoid impregnating a partner or avoid becoming pregnant, by practicing abstinence or using acceptable contraception

Exclusion Criteria:

* Has a baseline lower respiratory tract specimen Gram stain that shows the presence of Gram-positive cocci only
* Has confirmed or suspected community-acquired bacterial pneumonia (CABP)
* Has confirmed or suspected pneumonia of viral, fungal or parasitic origin
* Has HABP/VABP caused by an obstructive process, including lung cancer or other known obstruction
* Has a carcinoid tumor or carcinoid syndrome
* Has active immunosuppression defined as either receiving immunosuppressive medications or having a medical condition associated with immunodeficiency
* Is expected to survive for less than 72 hours
* Has a concurrent condition or infection that would preclude evaluation of therapeutic response
* Has received effective antibacterial drug therapy for the index infection of HABP/VABP for more than 24 hours continuously, during the previous 72 hours
* Has a history of serious allergy, hypersensitivity or a serious reaction to any penicillin or beta-lactamase inhibitors
* Female is pregnant, expecting to conceive, is breastfeeding or plans to breastfeed
* Has a history of seizure disorder requiring ongoing prior treatment with anti-convulsive therapy within the last 3 years
* Anticipates treatment with the following: valproic acid or divalproex sodium, serotonin re-uptake inhibitors, tricyclic antidepressants, or serotonin receptor antagonists, meperidine, buspirone, concomitant systemic antibacterial agents, antifungal or antiviral therapy for the index infection of HABP/VABP
* Is currently undergoing hemodialysis or peritoneal dialysis
* Is currently participating in, has participated in during the previous 30 days, or anticipates to participate in any other clinical study involving the administration of experimental medication
* Has previously participated in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 537 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Martin-Loeches I, Shorr AF, Kollef MH, Du J, Losada MC, Paschke A, DeRyke CA, Wong M, Jensen EH, Chen LF. Participant- and Disease-Related Factors as Independent Predictors of Treatment Outcomes in the RESTORE-IMI 2 Clinical Trial: A Multivariable Regression Analysis. Open Forum Infect Dis. 2023 May 4;10(6):ofad225. doi: 10.1093/ofid/ofad225. eCollection 2023 Jun. PMID 37383243
- [Derived] Patel M, Bellanti F, Daryani NM, Noormohamed N, Hilbert DW, Young K, Kulkarni P, Copalu W, Gheyas F, Rizk ML. Population pharmacokinetic/pharmacodynamic assessment of imipenem/cilastatin/relebactam in patients with hospital-acquired/ventilator-associated bacterial pneumonia. Clin Transl Sci. 2022 Feb;15(2):396-408. doi: 10.1111/cts.13158. Epub 2021 Oct 27. PMID 34704389
- [Derived] Titov I, Wunderink RG, Roquilly A, Rodriguez Gonzalez D, David-Wang A, Boucher HW, Kaye KS, Losada MC, Du J, Tipping R, Rizk ML, Patel M, Brown ML, Young K, Kartsonis NA, Butterton JR, Paschke A, Chen LF. A Randomized, Double-blind, Multicenter Trial Comparing Efficacy and Safety of Imipenem/Cilastatin/Relebactam Versus Piperacillin/Tazobactam in Adults With Hospital-acquired or Ventilator-associated Bacterial Pneumonia (RESTORE-IMI 2 Study). Clin Infect Dis. 2021 Dec 6;73(11):e4539-e4548. doi: 10.1093/cid/ciaa803. PMID 32785589

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult male and female participants requiring intravenous (IV) therapy for hospital-acquired bacterial pneumonia (HABP) or ventilator-assisted bacterial pneumonia (VABP) were recruited at 120 study centers in 28 countries.
Groups:
- IMI/REL: Participants received imipenem 500 mg + relebactam 250 mg + cilastatin 500 mg as a fixed dose combination (FDC) administered IV every 6 hours for a minimum of 7 days, up to 14 days. At the start of IMI/REL treatment, participants were treated empirically with 600 mg open-label linezolid administered IV every 12 hours until methicillin-resistant Staphylococcus aureus (MRSA) was ruled out. Participants with confirmed MRSA infection continued to receive 600 mg linezolid every 12 hours for a minimum of 7 days, up to 14 days total.
- PIP/TAZ: Participants received piperacillin 4000 mg + tazobactam 500 mg as a FDC administered IV every 6 hours for a minimum of 7 days, up to 14 days. At the start of PIP/TAZ treatment, participants were treated empirically with 600 mg open-label linezolid administered IV every 12 hours until MRSA was ruled out. Participants with confirmed MRSA infection continued to receive 600 mg linezolid every 12 hours for a minimum of 7 days, up to 14 days total.
Period: Overall Study
Arm/Group | IMI/REL | PIP/TAZ
Started | 268 | 269
Completed | 185 | 187
Not Completed | 83 | 82
Not completed — Adverse Event | 2 | 2
Not completed — Death | 44 | 58
Not completed — Lost to Follow-up | 2 | 1
Not completed — Protocol Violation | 6 | 7
Not completed — Physician Decision | 1 | 1
Not completed — Participant moved | 17 | 5
Not completed — Withdrawal parent/guardian | 0 | 1
Not completed — Withdrawal by Subject | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- IMI/REL: Participants received imipenem 500 mg + relebactam 250 mg + cilastatin 500 mg as a FDC administered IV every 6 hours for a minimum of 7 days, up to 14 days. At the start of IMI/REL treatment, participants were treated empirically with 600 mg open-label linezolid administered IV every 12 hours until MRSA was ruled out. Participants with confirmed MRSA infection continued to receive 600 mg linezolid every 12 hours for a minimum of 7 days, up to 14 days total.
- Total: Total of all reporting groups
Arm/Group | IMI/REL | PIP/TAZ | Total
Number analyzed (Participants) | 268 | 269 | 537
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.4 (17.0) | 58.9 (18.4) | 59.7 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 78 | 164
  Male | 182 | 191 | 373
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56 | 55 | 111
  Not Hispanic or Latino | 209 | 205 | 414
  Unknown or Not Reported | 3 | 9 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 8 | 13
  Asian | 42 | 37 | 79
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 6 | 10
  White | 208 | 209 | 417
  More than one race | 9 | 7 | 16
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With All-cause Mortality (ACM) Through Day 28 in the Modified Intention-to-treat (MITT) Population
Description: The percentage of participants in the MITT population with mortality due to any cause from randomization through Day 28 was determined for each arm.
Time Frame: Up to 28 days
Population: The MITT population includes all randomized participants who received ≥1 dose of study treatment and did not have only gram-positive cocci on Gram stain of the baseline lower respiratory tract (LRT) specimen.
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 264 | 267
Percentage of participants | 15.9 | 21.3
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Adjusted difference in all-cause mortality; Test type: Non-Inferiority — Non-inferiority was declared when the upper bound of the 2-sided 95% confidence interval (CI) for the difference in mortality (IMI/REL minus PIP/TAZ) was < 10 percentage points; p < 0.001, t-test, 1 sided; A one-sided alpha level of 0.025 was used to declare significance; Adjusted difference in ACM = -5.3, 95% CI 2-sided [-11.9 to 1.2] — Adjusted difference and 95% CI are based on the Miettinen & Nurminen method

2. Secondary Outcome: Percentage of Participants in the MITT Population With a Favorable Clinical Response (FCR) at Early Follow-up (EFU) Visit
Description: The percentage of participants with a FCR at EFU was determined for each arm. Favorable clinical response at EFU was defined as either "sustained cure" (all pre-therapy signs and symptoms of the index infection have resolved [or returned to "pre-infection status"] with no evidence of resurgence and no additional antibiotics are required) or "cure" (all pre-therapy signs and symptoms of the index infection have resolved [or returned to "pre-infection status"] and no additional antibiotics are required).
Time Frame: Up to 16 days after end of therapy (up to 30 days)
Population: The MITT population includes all randomized participants who received ≥1 dose of study treatment and did not have only gram-positive cocci on Gram stain of the baseline LRT specimen.
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 264 | 267
Percentage of participants | 61.0 | 55.8
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Adjusted difference in FCR; Test type: Non-Inferiority — Non-inferiority was declared when the lower bound of the 2-sided 95% CI for the difference in FCR (IMI/REL minus PIP/TAZ) was > 12.5 percentage points; p < 0.001, t-test, 1 sided; A one-sided alpha level of 0.025 was used to declare significance; Adjusted difference in FCR = 5.0, 95% CI 2-sided [-3.2 to 13.2] — Adjusted difference and 95% CI are based on the Miettinen & Nurminen method

3. Secondary Outcome: Percentage of Participants With ≥1 Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 30 days
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 266 | 269
Percentage of participants | 85.0 | 86.6
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Test type: Other — Difference in % with AE vs PIP/TAZ; Difference in % with AE = -1.7, 95% CI 2-sided [-7.7 to 4.3]

4. Secondary Outcome: Percentage of Participants Discontinuing Study Therapy Due to an AE
Description: as for outcome 3
Time Frame: Up to 14 days
Population: All participants who received ≥1 dose of study therapy are included.
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 266 | 269
Percentage of participants | 5.6 | 8.2
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Test type: Other — Difference in % discontinuing vs PIP/TAZ; Difference in % discontinuing = -2.5, 95% CI 2-sided [-7.1 to 1.8]

5. Secondary Outcome: Percentage of Participants With ACM in the Microbiological Modified Intention-to-treat (mMITT) Population
Description: The percentage of participants in the mMITT population with mortality due to any cause from randomization through Day 28 was determined for each arm.
Time Frame: Up to 28 days
Population: The mMITT population includes all randomized participants who received ≥1 dose of study treatment and did not have only gram-positive cocci only on baseline Gram stain and who have a baseline bacterial pathogen identified as the cause of HABP/VABP against which IMI/REL has been shown to have antibacterial activity.
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 215 | 218
Percentage of participants | 16.7 | 20.2
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Adjusted difference in all-cause mortality; Test type: Other; Adjusted difference in ACM = -3.5, 95% CI 2-sided [-10.9 to 3.6] — Adjusted difference and 95% CI are based on the Miettinen & Nurminen method

6. Secondary Outcome: Percentage of Participants With ACM at EFU in the MITT Population
Description: The percentage of participants in the MITT population with mortality due to any cause from randomization through EFU was determined for each arm.
Time Frame: Up to 16 days after end of therapy (up to 30 days)
Population: The MITT population includes all randomized participants who received ≥1 dose of study treatment and did not have only gram-positive cocci on Gram stain of the baseline specimen.
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 264 | 267
Percentage of participants | 14.8 | 19.5
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Adjusted difference in all-cause mortality; Test type: Non-Inferiority — Non-inferiority was declared when the upper bound of the 2-sided 95% CI for the difference in mortality (IMI/REL minus PIP/TAZ) was ≥ 10 percentage points; Adjusted difference in ACM = -4.6, 95% CI 2-sided [-11.0 to 1.7] — Adjusted difference and 95% CI are based on the Miettinen & Nurminen method

7. Secondary Outcome: Percentage of Participants With ACM at EFU in the mMITT Population
Description: The percentage of participants in the mMITT population with mortality due to any cause from randomization through EFU was determined for each arm.
Time Frame: Up to 16 days after end of therapy (up to 30 days)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 215 | 218
Percentage of participants | 15.3 | 18.3
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Adjusted difference in all-cause mortality; Test type: Other — Adjusted difference in ACM; Adjusted difference in ACM = -3.1, 95% CI 2-sided [-10.2 to 3.8] — Adjusted difference and 95% CI are based on the Miettinen & Nurminen method

8. Secondary Outcome: Percentage of Participants in the Clinically Evaluable (CE) Population With a FCR at On-therapy Visit 1 (OTX1) [Day 3]
Description: The percentage of participants with a FCR at OTX1 was determined for each arm. Favorable clinical response at OTX1 was defined as "improved" (majority of pre-therapy signs and symptoms of the index infection have improved or resolved [or returned to "pre-infection status"]).
Time Frame: Day 3 (OTX1)
Population: The CE population is all randomized participants with ≥1 dose of study therapy; had not only gram-positive cocci on baseline Gram stain; met important entry criteria; had no protocol deviations; received minimum duration of IV therapy; and have Day 3 clinical response data.
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 171 | 165
Percentage of participants | 70.8 | 72.8
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Adjusted difference in favorable clinical response; Test type: Other — Difference in FCR; Adjusted difference in FCR = -1.7, 95% CI 2-sided [-11.3 to 7.8] — Adjusted difference and 95% CI are based on the Miettinen & Nurminen method

9. Secondary Outcome: Percentage of Participants in the CE Population With a FCR at OTX2 (Day 6)
Description: The percentage of participants with a FCR at OTX2 was determined for each arm. Favorable clinical response at OTX2 was defined as "improved" (majority of pre-therapy signs and symptoms of the index infection have improved or resolved [or returned to "pre-infection status"]).
Time Frame: Day 6 (OTX2)
Population: The CE population is all randomized participants with ≥1 dose of study therapy; had not only gram-positive cocci on baseline Gram stain; met important entry criteria; had no protocol deviations; received minimum duration of IV therapy; and have Day 6 clinical response data.
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 171 | 165
Percentage of participants | 85.5 | 87.8
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Adjusted difference in favorable clinical response; Test type: Other — Difference in FCR; Adjusted difference in FCR = -2.2, 95% CI 2-sided [-9.8 to 5.5] — Adjusted difference and 95% CI are based on the Miettinen & Nurminen method

10. Secondary Outcome: Percentage of Participants in the CE Population With a FCR at OTX3 (Day 10)
Description: The percentage of participants with a FCR at OTX3 was determined for each arm. Favorable clinical response at OTX3 was defined as "improved" (majority of pre-therapy signs and symptoms of the index infection have improved or resolved [or returned to "pre-infection status"]).
Time Frame: Day 10 (OTX3)
Population: The CE population is all randomized participants with ≥1 dose of study therapy; had not only gram-positive cocci on baseline Gram stain; met important entry criteria; had no protocol deviations; received minimum duration of IV therapy; and have Day 10 clinical response data.
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 171 | 165
Percentage of participants | 89.6 | 83.6
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Adjusted difference in favorable clinical response; Test type: Other — Difference in favorable clinical response; Adjusted difference in FCR = 6.6, 95% CI 2-sided [-4.6 to 18.4] — Adjusted difference and 95% CI are based on the Miettinen & Nurminen method

11. Secondary Outcome: Percentage of Participants in the CE Population With a FCR at EOT Visit
Description: The percentage of participants with a FCR at EOT was determined for each arm. Favorable clinical response at EOT was defined as either "cure" (all pre-therapy signs and symptoms of the index infection have resolved [or returned to "pre-infection status"] and no additional antibiotics are required) or "improved" (the majority of pre-therapy signs and symptoms of the index infection have improved or resolved [or returned to "pre-infection status"] and no additional antibiotics are required).
Time Frame: From Day 7 to Day 14
Population: The CE population is all randomized participants with ≥1 dose of study therapy; had not only gram-positive cocci on baseline Gram stain; met important entry criteria; had no protocol deviations; received minimum duration of IV therapy; and have EOT clinical response data.
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 171 | 165
Percentage of participants | 84.7 | 85.3
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Adjusted difference in favorable clinical response; Test type: Other — Difference in FCR; Adjusted difference in FCR = -0.4, 95% CI 2-sided [-8.1 to 7.4] — Adjusted difference and 95% CI are based on the Miettinen & Nurminen method

12. Secondary Outcome: Percentage of Participants in the CE Population With a FCR at Day 28
Description: The percentage of participants with a FCR at Day 28 was determined for each arm. Favorable clinical response at Day 28 was defined as either "sustained cure" (all pre-therapy signs and symptoms of the index infection have resolved [or returned to "pre-infection status"] with no evidence of resurgence and no additional antibiotics are required) or "cure" (all pre-therapy signs and symptoms of the index infection have resolved [or returned to "pre-infection status"] and no additional antibiotics are required).
Time Frame: Day 28
Population: The CE population is all randomized participants with ≥1 dose of study therapy; had not only gram-positive cocci on baseline Gram stain; met important entry criteria; had no protocol deviations; received minimum duration of IV therapy; and have Day 28 clinical response data.
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 147 | 144
Percentage of participants | 70.5 | 75.6
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Adjusted difference in favorable clinical response; Test type: Other — Difference in FCR; Adjusted difference in FCR = -3.4, 95% CI 2-sided [-14.3 to 7.5] — Adjusted difference and 95% CI are based on the Miettinen & Nurminen method

13. Secondary Outcome: Percentage of Participants in the CE Population With a FCR at EFU Visit
Description: as for outcome 2
Time Frame: Up to 16 days after end of therapy (up to Day 30)
Population: The CE population is all randomized participants with ≥1 dose of study therapy; had not only gram-positive cocci on baseline Gram stain; met important entry criteria; had no protocol deviations; received minimum duration of IV therapy; and have EFU clinical response data.
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 147 | 144
Percentage of participants | 74.3 | 79.4
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Adjusted difference in favorable clinical response; Test type: Other — Difference in FCR; Adjusted difference in FCR = -3.7, 95% CI 2-sided [-13.6 to 6.4] — Adjusted difference and 95% CI are based on the Miettinen & Nurminen method

14. Secondary Outcome: Percentage of Participants in the MITT Population With a FCR at OTX1 (Day 3)
Description: as for outcome 8
Time Frame: Day 3 (OTX1)
Population: The MITT population includes all randomized participants who received ≥1 dose of study treatment, did not have only gram-positive cocci on Gram stain of the baseline specimen, and have Day 3 data.
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 264 | 267
Percentage of participants | 68.0 | 64.7
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Adjusted difference in favorable clinical response; Test type: Other — Difference in FCR; Adjusted difference in FCR = 3.5, 95% CI 2-sided [-4.6 to 11.6] — Adjusted difference and 95% CI are based on the Miettinen & Nurminen method

15. Secondary Outcome: Percentage of Participants in the MITT Population With a FCR at OTX2 (Day 6)
Description: as for outcome 9
Time Frame: Day 6 (OTX2)
Population: The MITT population includes all randomized participants who received ≥1 dose of study treatment, did not have only gram-positive cocci on Gram stain of the baseline specimen, and have Day 6 data.
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 264 | 267
Percentage of participants | 83.5 | 83.1
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Adjusted difference in favorable clinical response; Test type: Other — Difference in FCR; Adjusted difference in FCR = 0.5, 95% CI 2-sided [-6.3 to 7.4] — Adjusted difference and 95% CI are based on the Miettinen & Nurminen method

16. Secondary Outcome: Percentage of Participants in the MITT Population With a FCR at OTX3 (Day 10)
Description: as for outcome 10
Time Frame: Day 10 (OTX3)
Population: The MITT population includes all randomized participants who received ≥1 dose of study treatment, did not have only gram-positive cocci on Gram stain of the baseline specimen, and have Day 10 data.
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 264 | 267
Percentage of participants | 83.5 | 80.4
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Adjusted difference in favorable clinical response; Test type: Other — Difference in FCR; Adjusted difference in FCR = 3.4, 95% CI 2-sided [-7.1 to 14.2] — Adjusted difference and 95% CI are based on the Miettinen & Nurminen method

17. Secondary Outcome: Percentage of Participants in the MITT Population With a FCR at EOT
Description: as for outcome 11
Time Frame: From Day 7 to Day 14
Population: The MITT population includes all randomized participants who received ≥1 dose of study treatment, did not have only gram-positive cocci on Gram stain of the baseline specimen, and have EOT data.
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 264 | 267
Percentage of participants | 74.2 | 69.7
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Adjusted difference in favorable clinical response; Test type: Other — Difference in FCR; Adjusted difference in FCR = 4.4, 95% CI 2-sided [-3.1 to 12.0] — Adjusted difference and 95% CI are based on the Miettinen & Nurminen method

18. Secondary Outcome: Percentage of Participants in the MITT Population With a FCR at Day 28
Description: as for outcome 12
Time Frame: Day 28
Population: The MITT population includes all randomized participants who received ≥1 dose of study treatment, did not have only gram-positive cocci on Gram stain of the baseline specimen, and have Day 28 data.
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 264 | 267
Percentage of participants | 51.9 | 50.6
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Adjusted difference in favorable clinical response; Test type: Other — Difference in FCR; Adjusted difference in FCR = 1.1, 95% CI 2-sided [-7.2 to 9.4] — Adjusted difference and 95% CI are based on the Miettinen & Nurminen method

19. Secondary Outcome: Percentage of Participants in the mMITT Population With a Favorable Microbiological Response (FMR) at End of Treatment (EOT) Visit
Description: The percentage of participants with a FMR at EOT was determined for each arm. Favorable microbiological response at EOT was defined as either "eradication" (a lower respiratory tract culture taken at EOT showing eradication of baseline pathogen) or "presumed eradication" (no specimen collected because the participant deemed clinically cured or improved).
Time Frame: From Day 7 to Day 14
Population: The mMITT population includes all randomized participants who received ≥1 dose of study treatment, did not have only gram-positive cocci only on baseline Gram stain, have a baseline bacterial pathogen identified as the cause of HABP/VABP against which IMI/REL has been shown to have antibacterial activity, and have EOT data.
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 215 | 218
Percentage of participants | 77.2 | 67.9
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Adjusted difference in favorable microbiological response; Test type: Other — Difference in FMR; Adjusted difference in FMR = 9.7, 95% CI 2-sided [1.6 to 17.9] — Adjusted difference and 95% CI are based on the Miettinen & Nurminen method

20. Secondary Outcome: Percentage of Participants in the mMITT Population With a FMR at EFU Visit
Description: The percentage of participants with a FMR at EFU was determined for each arm. Favorable microbiological response at EOT was defined as either "eradication" (a lower respiratory tract culture taken at EFU showing eradication of baseline pathogen) or "presumed eradication" (no specimen collected because the participant deemed clinically cured or improved).
Time Frame: Up to 16 days after end of therapy (up to Day 30)
Population: The mMITT population includes all randomized participants who received ≥1 dose of study treatment, did not have only gram-positive cocci only on baseline Gram stain, have a baseline bacterial pathogen identified as the cause of HABP/VABP against which IMI/REL has been shown to have antibacterial activity, and have EFU data.
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 215 | 218
Percentage of participants | 67.9 | 61.9
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Adjusted difference in favorable microbiological response; Test type: Other — Difference in FMR; Adjusted difference in FMR = 6.2, 95% CI 2-sided [-2.7 to 15.0] — Adjusted difference and 95% CI are based on the Miettinen & Nurminen method

21. Secondary Outcome: Percentage of Participants in the Microbiologically Evaluable (ME) Population With a FMR at EOT Visit
Description: as for outcome 19
Time Frame: From Day 7 to Day 14
Population: The ME population is all randomized participants with ≥1 dose of study therapy; not only gram-positive cocci on baseline Gram stain; IMI/REL-sensitive baseline pathogen as cause of HABP/VABP; met entry criteria; no protocol deviations; received minimum duration of IV therapy; have microbiological EOT data and LRT culture available.
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 140 | 133
Percentage of participants | 87.1 | 85.5
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Adjusted difference in favorable microbiological response; Test type: Other — Difference in FMR; Adjusted difference in FMR = 2.5, 95% CI 2-sided [-5.5 to 11.0] — Adjusted difference and 95% CI are based on the Miettinen & Nurminen method

22. Secondary Outcome: Percentage of Participants in the ME Population With a FMR at EFU Visit
Description: as for outcome 19
Time Frame: Up to 16 days after end of therapy (up to Day 30)
Population: The ME population is all randomized participants with ≥1 dose of study therapy; not only gram-positive cocci on baseline Gram stain; IMI/REL-sensitive baseline pathogen as cause of HABP/VABP; met entry criteria; no protocol deviations; received minimum duration of IV therapy; have microbiological EFU data and LRT culture available.
Measure: Number; unit: Percentage of participants
Arm/Group | IMI/REL | PIP/TAZ
Number analyzed (Participants) | 121 | 117
Percentage of participants | 89.9 | 86.4
Statistical Analysis 1: Comparison: IMI/REL vs PIP/TAZ; Adjusted difference in favorable microbiological response; Test type: Other — Difference in FMR; Adjusted difference in FMR = 4.7, 95% CI 2-sided [-4.0 to 14.1] — Adjusted difference and 95% CI are based on the Miettinen & Nurminen method

ADVERSE EVENTS:
Time Frame: Up to 30 days
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. All randomized participants who received ≥1 dose of IV study therapy are included in the analysis.
Arm/Group | IMI/REL | PIP/TAZ
All-Cause Mortality (participants affected / at risk) | 44/266 | 58/269
Serious Adverse Events (participants affected / at risk) | 71/266 | 86/269
Other Adverse Events (participants affected / at risk) | 98/266 | 105/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMI/REL (N=266) | PIP/TAZ (N=269)
Splenic lesion (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 10 (12) | 7 (9)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 2 (2) | 2 (2)
Cardiovascular insufficiency (Cardiac disorders) | 3 (3) | 4 (4)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Brain death (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 6 (6)
Vascular stent thrombosis (General disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 2 (2)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Brain abscess (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Carbuncle (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Fungaemia (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 1 (1)
Meningitis (Infections and infestations) | 1 (1) | 1 (1)
Neurological infection (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 3 (3)
Pneumonia acinetobacter (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Post procedural sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 3 (3)
Septic shock (Infections and infestations) | 7 (7) | 4 (4)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Spinal cord infection (Infections and infestations) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Implant tissue necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal shock (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Wound evisceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Basilar artery thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Brain dislocation syndrome (Nervous system disorders) | 1 (1) | 3 (3)
Brain oedema (Nervous system disorders) | 0 (0) | 3 (3)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 3 (3)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (2)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 8 (8)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 3 (3) | 2 (2)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Haemodynamic instability (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMI/REL (N=266) | PIP/TAZ (N=269)
Anaemia (Blood and lymphatic system disorders) | 28 (30) | 27 (28)
Diarrhoea (Gastrointestinal disorders) | 21 (22) | 29 (32)
Pyrexia (General disorders) | 11 (19) | 20 (29)
Alanine aminotransferase increased (Investigations) | 23 (25) | 18 (18)
Aspartate aminotransferase increased (Investigations) | 29 (31) | 19 (19)
Hypokalaemia (Metabolism and nutrition disorders) | 18 (19) | 24 (25)
Hyponatraemia (Metabolism and nutrition disorders) | 14 (15) | 3 (3)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 14 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT02493764/Prot_SAP_000.pdf